CLINICAL TRIAL: NCT00264355
Title: Metabolic Pattern of Cyclosporine A - Association of Secondary- and Cyclic Metabolites With Acute Renal Failure in Heart Transplant Recipients
Brief Title: Metabolic Pattern of Cyclosporine A and Acute Renal Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HeartTx-ARF
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2007-09-06 (Estimated); Status verified 2007-09

CONDITIONS: Heart Transplantation; Acute Renal Failure
Keywords: cyclosporine; metabolites; metabolic pattern; genotypes
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cyclosporine

INTERVENTIONS:
Drug: cyclosporine A

SUMMARY:
Following heart transplantation many patients develop acute renal failure in the early posttransplant phase and some are in need of renal replacement therapy for shorter or longer time. The cause of this acute renal failure is most probably multi factorial but many reports indicate that cyclosporine has a central role in the pathophysiology and it is generally recommended to lower the cyclosporine load to patients developing acute renal failure in this population.

Several in vitro studies on renal cells in culture indicate that the primary metabolites of cyclosporine (AM1, AM9, AM4N) are less toxic to the kidney than cyclosporine itself. However, the secondary metabolite AM19 as well as the cyclic metabolites AM1c and AM1c9 has been associated with decreased renal function and nephrotoxicity renal transplant recipients.

The primary objective of this pilot study is to investigate if the concentrations of secondary- and cyclic metabolites of cyclosporine (AM19, AM1c, AM1c9) is related to development of acute renal failure in the early posttransplant phase following heart transplantation.

Secondary objectives are to investigate associations between genotypes of P-glycoprotein and CYP3A5 and the metabolic pattern of cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant recipients receiving CsA as part of their immunosuppressive therapy.
* 18 years of age or older.
* Signed informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary analysis of cyclosporine and metabolite concentrations and ratios will be compared between the patients developing acute renal failure and those who do not

SECONDARY OUTCOMES:
Regression analysis comparing concentrations/ratios and actual renal function (continuously parameter)
Descriptive listing of cyclosporine and metabolites concentrations in CYP3A5*3/*3 patients compared to the other patients. It is anticipated that an exploratory analysis will be performed to compare the two groups.
Descriptive listing of CsA and metabolites concentrations in patients with different combinations of MDR-1 genotypes compared to the other patients. It is anticipated that an exploratory analysis will be performed to compare the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, Ph.D., Study Director — University of Oslo School of Pharmacy; Arnt Fiane, MD, Ph.D., Principal Investigator — Rikshospitalet, Department of Thoracic surgery
Locations (1):
- Rikshospitalet, Department of Thoracic surgery, Oslo, Norway